CLINICAL TRIAL: NCT00568867
Title: Evaluation of Preexisting Immunity Markers in Human Tumor Tissue Sample
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Jeffrey A. Norton, Stanford University School of Medicine
Other Study IDs: SU-11072007-830; 97310 (Other: Stanford University Alternate IRB Approval Number); VAR0018 (Other: Stanford University); NCT00507624 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate markers of immune response in human tumor samples.

DETAILED DESCRIPTION:
Cancer immunotherapy has been shown to be effective in isolated instances, but ineffective in most patients. The reason for this inconsistency, and the conditions necessary for successful immunotherapy, are not well understood. Our studies in animal tumor models indicate that the effectiveness of IL-12-based immunotherapy depends upon the presence of a preexisting immune response to the tumor. The presence of T cell infiltrates and IFN-gamma expression in tumor indicate such an immune response. We therefore plan to evaluate the existing immune response in human tumor samples in an effort to identify those patients most likely to respond to therapy with IL-12.

ELIGIBILITY:
Inclusion Criteria:Any adult patient with a tumor who is scheduled to undergo surgery to either remove or biopsy the tumor. Exclusion Criteria:Patients without tumor and pediatric patients (children) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient with a tumor who is scheduled to undergo surgery to either remove or biopsy the tumor.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Norton, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States